CLINICAL TRIAL: NCT02959905
Title: Phase I Clinical Trial of TSA-CTL (Tumor Specific Antigen-Induced Cytotoxic T Lymphocytes) In the Treatment of Advanced Solid Tumors
Brief Title: Treatment of Advanced Solid Tumors With TSA-CTL(Tumor Specific Antigen-Induced Cytotoxic T Lymphocytes)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BGI, China (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGI-001; 2016-FXY-040 (Other Grant/Funding Number: Institutional Review Board of Sun Yat-Sen University); B2016-039 (Other Grant/Funding Number: ethics committee of Sun Yat-Sen University)
Record Dates: First submitted 2016-10-21; First posted 2016-11-09 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Solid Cancer
Keywords: Metastatic Melanoma; Colorectal Cancer; neoantigen
MeSH Terms: conditions — Melanoma; Colorectal Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- medium-dose lymphodepletion regimen (Experimental): Patients will receive medium-dose lymphodepletion regimen consisting of cyclophosphamide and fludarabine followed by TSA-CTL.
  Interventions: Biological: TSA-CTL; Drug: Fludarabine; Drug: Cyclophosphamide
- low-dose lymphodepletion regimen (Experimental): Patients will receive low-dose lymphodepletion regimen consisting of cyclophosphamide and fludarabine followed by TSA-CTL.
  Interventions: Biological: TSA-CTL; Drug: Cyclophosphamide; Drug: Fludarabine
- No lymphodepletion regimen (Experimental): Patients will only receive TSA-CTL.
  Interventions: Biological: TSA-CTL

INTERVENTIONS:
Biological: TSA-CTL — Patients will receive TSA-CTL iv over 20-30 minutes on day 0.
  Other Names: Tumor Specific Antigen Induced Cytotoxic Lymphocyte
Drug: Cyclophosphamide — Cyclophosphamide 500 mg/m2/day iv on day -5 for one day.
  Other Names: Cytoxan
  Arms: low-dose lymphodepletion regimen
Drug: Fludarabine — Fludarabine 25 mg/m2/day iv over 30 minutes on day -5 and -4 for two days.
  Other Names: Fludarabine Phosphate
  Arms: low-dose lymphodepletion regimen; medium-dose lymphodepletion regimen
Drug: Cyclophosphamide — Cyclophosphamide 500 mg/m2/day iv on day -5 and -4 for two days.
  Other Names: Cytoxan
  Arms: medium-dose lymphodepletion regimen

SUMMARY:
The primary objective of this study is to evaluate the safety of TSA-CTL in the treatment of advanced solid tumors.

The secondary objective of this study is to evaluate preliminarily the effect of TSA-CTL in the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This is a single arm, open label and non-randomized clinical study with two parts.

In Part 1, 9 subjects with advanced solid tumors will be enrolled into Groups A (no non-myeloablative lymphodepletion), B and C (non-myeloablative lymphodepletion with different chemotherapy intensities) to assess the safety and dose intensity of non-myeloablative lymphodepletion chemotherapy before cell infusion.

Depending on results in Part 1, the study may proceed to Part 2, where 15 subjects with advanced solid tumors will be enrolled to receive TSA-CTL cell infusions with or without non-myeloablative lymphodepletion.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years of age and less than or equal to 70 years of age; all genders.
2. Advanced solid tumors including but not limited to some high frequency somatic mutations, such as melanoma, colorectal cancer, gastric cancer, esophageal cancer, squamous cell carcinoma of the lung, triple-negative breast cancer, etc.
3. Advanced solid tumors patients who are HLA - A0201 /A1101/A2402 subtypes.
4. Measurable solid tumors with at least one lesion that is resectable or tumor biopsies for DNA extraction.
5. Patients who failed or were intolerant to standard treatment.
6. Patients (or their legal representatives) who are able to understand and sign the Informed Consent Form and willing to sign a durable power of attorney.
7. Clinical performance status of ECOG is 0 or 1 and expected lifetime is greater than six month and patients who are able to cooperate to observe adverse reactions and the effect of the treatment.
8. Patients of both genders must be willing to practice birth control from the time of enrollment to five months after treatment on this study.
9. Serology: HIV antibody(-), hepatitis B antigen(-), and hepatitis C antibody(-). A fertile woman must have a negative pregnancy test. Hematology: Absolute neutrophil count is greater than 1500/mm3 without the support of filgrastim; WBC is greater than or equal to 3000/mm3; lymphocyte count is greater than or equal to 800/mm3; Platelet count is greater than or equal to 100,000/mm3; Hemoglobin is greater than or equal to 9.0 g/dL ; Chemistry: Serum ALT/AST is less than or equal to 2.5 times the upper limit of normal; Serum Creatinine is less than or equal to 1.5 times the upper limit of normal ; Total bilirubin is less than or equal to 1.5 the upper limit of normal, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 times the upper limit of normal.
10. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the lymphodepletion regimen, and toxicities must have recovered to grade 1 or less (except for toxicities such as alopecia or vitiligo).

Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Any primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
3. Opportunistic infection.
4. History of autoimmune disease.
5. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system.
6. Systemic steroid therapy in the past 4 weeks.
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. Patients with unstable brain metastases.
9. Choroidal melanoma and clear cell sarcoma patients.
10. Negative for expression of MHC molecules.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v5.0. | one month
  Keep records the adverse events experienced by subjects in 30 days after the first infusion.

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | one year
  DCR is defined as the proportion of participants with tumor size reduction(CR,PR) and stable disease(SD) assessed by RECIST 1.1 and iRECIST.
overall survival(OS) | one year
  The time from the first infusion of Investigational Product until death.
progression-free survival(PFS) | one year
  PFS is defined as the time from the first infusion of Investigational Product until objective tumor progression, as assessed by RECIST 1.1 and iRECIST, or death, whichever occurs first.
Duration of Response(DOR) | one year
  DOR refers to the period from the first evaluation of tumor as CR or PR to the first evaluation as PD(Progressive Disease) per RECIST1.1 and iRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Sh Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403
- [Result] Carreno BM, Magrini V, Becker-Hapak M, Kaabinejadian S, Hundal J, Petti AA, Ly A, Lie WR, Hildebrand WH, Mardis ER, Linette GP. Cancer immunotherapy. A dendritic cell vaccine increases the breadth and diversity of melanoma neoantigen-specific T cells. Science. 2015 May 15;348(6236):803-8. doi: 10.1126/science.aaa3828. Epub 2015 Apr 2. PMID 25837513
- [Result] Prickett TD, Crystal JS, Cohen CJ, Pasetto A, Parkhurst MR, Gartner JJ, Yao X, Wang R, Gros A, Li YF, El-Gamil M, Trebska-McGowan K, Rosenberg SA, Robbins PF. Durable Complete Response from Metastatic Melanoma after Transfer of Autologous T Cells Recognizing 10 Mutated Tumor Antigens. Cancer Immunol Res. 2016 Aug;4(8):669-78. doi: 10.1158/2326-6066.CIR-15-0215. Epub 2016 Jun 16. PMID 27312342
- [Derived] Li D, Chen C, Li J, Yue J, Ding Y, Wang H, Liang Z, Zhang L, Qiu S, Liu G, Gao Y, Huang Y, Li D, Zhang R, Liu W, Wen X, Li B, Zhang X, Zhang X, Xu RH. A pilot study of lymphodepletion intensity for peripheral blood mononuclear cell-derived neoantigen-specific CD8 + T cell therapy in patients with advanced solid tumors. Nat Commun. 2023 Jun 10;14(1):3447. doi: 10.1038/s41467-023-39225-7. PMID 37301885